CLINICAL TRIAL: NCT05025852
Title: A Multi-centre Follow up Study of the Effect of In-utero Exposure to Metformin in 5-11 Year Old Offspring of Mothers in the MiTy Trial
Brief Title: The Effect of In-utero Exposure to Metformin in 5-11 Year Old Offspring of Mothers in the MiTy Trial
Acronym: MiTy Tykes
Status: Recruiting | Type: Observational
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Sunnybrook Research Institute (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: CTO 3632
Record Dates: First submitted 2021-08-11; First posted 2021-08-27 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Mellitus, Type 2; Pregnancy in Diabetic; Child Obesity; Child Development
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Pregnancy in Diabetics; Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — A blood sample will be taken to be analyzed for markers of metabolic syndrome.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Metformin exposed in utero: Offspring of mothers who were exposed to metformin during pregnancy in the MiTy trial.
- Placebo exposed in utero: Offspring of mothers who were not exposed to metformin during pregnancy in the MiTy trial.

SUMMARY:
The incidence of diabetes in pregnancy is rising, with rates of 1 in 7 pregnancies globally. Metformin is used for type 2 diabetes (T2DM) outside of pregnancy and is now increasingly prescribed during pregnancy. There are some concerns as metformin crosses the placenta and effects on offspring exposed during pregnancy are unknown. Animal and human evidence indicate that metformin may create an atypical in-utero environment similar to under-nutrition which has been associated with adult obesity. This is supported by studies in children of mothers treated with metformin in other populations where an increase in childhood obesity was found at 4-9 years of age. We now have evidence from the MiTy trial, that offspring of metformin-exposed women with T2DM have less large infants and are less adipose at birth, but are also more likely to be small for gestational age (SGA). These effects could lead to benefit or harm in the long-term. Offspring of MiTy mothers are currently being followed up to 2 years. Given that long-term effects may not be evident until 5 years of age, it is imperative to follow these children longer.

Goals/Research Aims:To determine whether in-utero exposure to metformin, in offspring of women with T2DM, is beneficial or harmful in the long-term.

Research Questions: 1. In offspring of women with T2DM, how does treatment with metformin during pregnancy affect a) adiposity b) growth over time c) metabolic syndrome d) cognitive and behavioral measures:2. What factors predict altered childhood adiposity and insulin resistance in these offspring?

Primary Outcome: Body mass index (BMI) z-score.

Secondary Outcomes: 1) other measures of adiposity (i.e. skinfolds, 2) growth over time 3) measures of insulin resistance 4) adipocytokines 5)neurodevelopment

Expected Outcomes Given these increasing concerns, this study will inform the best treatment for pregnant mothers with diabetes by studying the long-term outcomes of children exposed to metformin during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Liveborn offspring of women who participated in the MiTy trial.

Exclusion Criteria:

* Offspring with major congenital anomalies that would affect growth or development (these children have already been excluded from MiTy Kids).

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Offspring of women with type 2 diabetes who participated in the MiTy trial will be recruited for participation.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index (BMI) z-score | 5-11 years of age
  Using WHO or other appropriate growth charts

SECONDARY OUTCOMES:
Skinfold measurements | 5-11 years of age
  triceps, subscapular and suprailiac skinfold thicknesses
Sum of skinfold measurements: | 5-11 years of age
  sum of triceps, subscapular and suprailiac skinfold thicknesses
Triceps skinfolds z-scores | 5-11 years of age
  Using WHO or other appropriate growth charts
Ratio of the central to peripheral skinfold ratio | 5-11 years of age
  ratio of the central (suprailiac) to peripheral (triceps) skinfold ratio;
Overweight and obesity status | 5-11 years of age
  Defined using WHO or other appropriate growth charts
Waist circumference | 5-11 years of age
  Waist circumference measurement
Waist to height ratio | 5-11 years of age
  Waist and height measurements
Growth trajectory | 5-11 years of age
  Longitudinal growth outcomes will be assessed using adiposity measurements from the MiTy trial (newborns) and at 3, 6, 12, 18 and 24 months from the MiTy Kids trial, to ages 5-11 years in the MiTy Tykes trial.
Fat mass | 5-11 years of age
  Using the Tanita SC-240 bioimpedance analyzer (BIA)
Percentage of body fat | 5-11 years of age
  Using the Tanita SC-240 bioimpedance analyzer (BIA)
Measures of insulin resistance and metabolic syndrome | 5-11 years of age
  The following measurements combined will contribute to the assessment of insulin resistance and metabolic syndrome: fasting glucose, fasting insulin, fasting insulin-to-glucose ratio, and the HOMA-IR, serum levels of leptin, adiponectin and lipids
Neurocognitive development | 5-11 years of age
  Attention Deficit Hyperactivity Disorder (ADHD)-5 Rating scale
Neurocognitive development | 5-11 years of age
  Children's Communication Checklist (CCC-2)
Neurocognitive development | 5-11 years of age
  Social Responsiveness Scale (SRS-2)

CONTACTS AND LOCATIONS:
Overall Officials: Denice Feig, MD, Principal Investigator — Mount Sinai Hospital, Toronto, ON, Canada
Locations (12):
- Australia (2):
  - Campbelltown Hospital, Campbelltown, New South Wales
  - Mater Misericordiae, Brisbane, Queensland
- Canada (10):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Children's Health Research Institute of Manitoba (CHRIM), Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - St Joseph's Health Care, London, Ontario
  - The Scarborough Hospital, Scarborough Village, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Hospital Maisonneuve-Rosemont, Montreal, Quebec
  - Chuq-Chul, Québec, Quebec